CLINICAL TRIAL: NCT04227184
Title: Investigation of Brain Mechanisms Involved in Urgency Urinary Incontinence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Becky Clarkson (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Becky Clarkson, Research Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: STUDY19090167; R01AG064251 (NIH)
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Urgency Urinary Incontinence
Keywords: Urinary Incontinence; Urgency urinary incontinence; Trospium
MeSH Terms: conditions — Urinary Incontinence | interventions — trospium chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo/Trospium (Experimental): Placebo first for 12 weeks followed by Trospium for 12 weeks.
  Interventions: Drug: Trospium; Drug: Placebo oral tablet
- Trospium/Placebo (Experimental): Trospium first for 12 weeks followed by Placebo for 12 weeks
  Interventions: Drug: Trospium; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Trospium — Drug to treat overactive bladder
  Other Names: Sanctura
Drug: Placebo oral tablet — Placebo tablet containing no active drug
  Other Names: Placebo

SUMMARY:
This is a randomized double-blind crossover trial of trospium and placebo in women with urgency urinary incontinence, with evaluation (history, physical, incontinence evaluation and brain MRI) at baseline, and after each course of therapy. The investigators will evaluate functional brain changes in relation to bladder improvement in order to improve our knowledge of the brain's role in the continence mechanism.

DETAILED DESCRIPTION:
Urgency urinary incontinence (UUI) costs the US $83 billion/year, owing in large part to its increased prevalence with age, particularly in women: 9% of those over age 18 and 36% of those over age 65. UUI also impairs quality of life, social interaction, and independence; contributes to functional decline; and increases risk for falls, hip fractures, UTIs, urosepsis, anxiety, depression, and institutionalization.The cause of UUI is unknown. Its urgency and leakage are usually ascribed to detrusor overactivity (DO, involuntary detrusor contraction), suggesting that the cause is intrinsic to the bladder even though DO is not always confirmed on testing. Because of this assumption, most therapies target the bladder albeit with only moderate success: e.g., anticholinergics reduce incontinence episodes but their benefit and tolerability (especially for older adults) are sufficiently low that 75% of patients discontinue them within a year. By contrast, therapies such as biofeedback-assisted pelvic muscle therapy (BFB) tackle behaviors. Moreover, the use of biofeedback to retrain the brain shows that the central control mechanism can be targeted and improved. Thus, the present proposal is designed to further elucidate this mechanism, thereby paving the way for discovery of new and more effective ways to control UUI. These could transform current treatment and either complement or supplant current therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 60+ years old
2. Has UUI or urge-predominant mixed incontinence at least 5 times/ week for > 3 months despite treatment for reversible causes

Exclusion Criteria:

1. conditions/medications contraindicating trospium
2. If currently taking anticholinergic medications (participant must refrain from anticholinergic medications for 4 weeks prior enrollment in order to be eligible)
3. Impaired mobility or cognition sufficient to preclude following study procedures; MoCA test score <24/30; a clinically-apparent neurological condition
4. Prolapse beyond the hymen
5. Interstitial cystitis
6. Spinal cord injury
7. History of pelvic radiation or advanced uterine/bladder cancer
8. Urethral obstruction (uroflow); PVR >200 ml
9. Medical instability
10. Prior UUI treatment with onabotulinum toxin or neuromodulation
11. Drug interaction or expected medication change during the study
12. Conditions requiring IV antibacterial prophylaxis
13. New incontinence treatment < 3 months prior to enrollment
14. Fecal incontinence, and symptomatic colitis/IBS
15. Contraindications to MRI.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Potential participants must be biologically female
Enrollment: 207 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Structural brain changes | Baseline to 12 weeks
  Change in grey and white matter volume on MRI compared between responders and non-responders to therapy/placebo. Grey matter and white matter volume of important brain structures will be compared, along with structural integrity of white matter pathways via tractography.
Structural brain changes | 12 to 24 weeks
  Change in grey and white matter volume on MRI compared between responders and non-responders to therapy/placebo. Grey matter and white matter volume of important brain structures will be compared, along with structural integrity of white matter pathways via tractography.
Functional brain changes | Baseline to 12 weeks
  Change in brain functional response to an infusion/withdrawal protocol compared between responders and non-responders to therapy/placebo. Changes are displayed as a map of t-values for each voxel of the brain, showing likelihood of statistical significance of changes.
Functional brain changes | 12 to 24 weeks
  Change in brain functional response to an infusion/withdrawal protocol compared between responders and non-responders to therapy/placebo. Changes are displayed as a map of t-values for each voxel of the brain, showing likelihood of statistical significance of changes.

CONTACTS AND LOCATIONS:
Overall Officials: Becky Clarkson, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification may be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following publication, no end date
Access Criteria: Any purpose

DOCUMENTS (1):
  • Informed Consent Form (2025-04-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT04227184/ICF_000.pdf